CLINICAL TRIAL: NCT06897839
Title: Randomized, Double-Blind Parallel-Group, Adaptive, Three-Arm, Phase 2b/3 Multicenter Study to Evaluate the Efficacy and Safety of Zelpultide Alfa in Preventing Bronchopulmonary Dysplasia (BPD) in High-Risk Preterm Neonates Compared to Standard of Care (SOC)
Brief Title: Efficacy and Safety of Zelpultide Alfa in Preterm Neonates at High Risk of Developing Bronchopulmonary Dysplasia (BPD)
Acronym: ZELA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Airway Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZEL-003; 2024-513420-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-20; First posted 2025-03-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: BPD; Zelpultide alfa; AT-100
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Zelpultide alfa 4 mg/kg plus standard of care (Experimental): In addition to the preterm neonate standard of care, the subjects randomized to this treatment arm will receive up to 7 administrations of zelpultide alfa at 4 mg/kg (birth weight) in 24 h intervals while the subjects are still intubated.
  Interventions: Drug: Zelpultide alfa
- Placebo (air-sham) plus standard of care (Sham Comparator): In addition to the preterm neonate standard of care, approximately 1 mL of air drawn into a dosing syringe will be administered up to 7 times to neonate subjects randomized to the control (placebo) arm, following the same means and intervals as in the treatment arm.
  Interventions: Other: Air-sham
- Zelpultide alfa 6 mg/kg plus standard of care (Experimental): In addition to the preterm neonate standard of care, the subjects randomized to this treatment arm will receive up to 7 administrations of zelpultide alfa at 6 mg/kg (birth weight) in 24 h intervals while the subjects are still intubated.
  Interventions: Drug: Zelpultide alfa

INTERVENTIONS:
Other: Air-sham — Room air for intratracheal administration
  Arms: Placebo (air-sham) plus standard of care
Drug: Zelpultide alfa — Reconstituted Zelpultide alfa for intratracheal administration
  Other Names: AT-100; rhSP-D
  Arms: Zelpultide alfa 4 mg/kg plus standard of care; Zelpultide alfa 6 mg/kg plus standard of care

SUMMARY:
This is a randomized, parallel-group, double-blind, placebo-controlled multicenter phase 2b/3 study with an adaptive seamless design.

The goal fo this study is to determine if an investigational drug, Zelpultide Alfa, can reduce the occurrence of Bronchopulmonary Dysplasia (BPD) in extremely premature babies.

The study comprises 2 parts:

* Part 1: Phase 2b, dose selection and exploratory efficacy and safety.
* Part 2: Phase 3, confirmatory efficacy and safety.

In Part 1, the study subjects will be randomized with a 1:1:1 allocation ratio to either :

1. Standard of care + zelpultide alfa 4 mg/kg or,
2. Standard of care + zelpultide alfa 6 mg/kg or,
3. Standard of care + placebo (air-sham).

In Part 1, all three arms will be evaluated descriptively to support dose selection based on safety, tolerability, and exploratory efficacy signals. Upon completion of Part 1, the DSMC will recommend which Phase 2b dose ("selected dose") to progress into Part 2 to the Study Steering Committee, which will decide the dose for Part 2 (Phase 3). A sample size reassessment will be performed after Part 1 completion.

In Part 2, the selected dose of zelpultide alfa will be compared against placebo (air-sham) in a confirmatory analysis on the primary and key secondary endpoints. The study subjects will be randomized with a 1:1 allocation ratio to either:

1. Standard of care + zelpultide alfa (selected dose from Part 1), or
2. Standard of care + placebo (air-sham). The main objective in part 2 is to compare the efficacy of zelpultide alfa added to standard of care versus standard of care plus placebo (air-sham) in terms of incidence of grade 2 and grade 3 bronchopulmonary dysplasia (BPD) and death in neonates at high risk for developing BPD.

In both parts, treatment will be administered intratracheally. Participants will receive up to 7 administrations of zelpultide alfa at (4mg/kg or 6 mg/kg) or air-sham in 24 h intervals while the subjects are still intubated per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Born between gestational age (GA) 22 0/7 to 27 6/7 weeks, inclusive.
2. Received at least 1 dose of SOC-indicated animal-derived pulmonary surfactant treatment after birth.
3. Intubated and on invasive mechanical ventilation per SOC.
4. Able to receive the first dose of zelpultide alfa or air-sham at least 15 min after the surfactant administration but within 96 h of birth and within 48 h from the start of invasive mechanical ventilation. Subjects extubated and re-intubated after their pulmonary surfactant dose(s) are eligible as long as the inclusion criteria are met.
5. Informed consent and personal information authorization form signed by the subject's parent(s) or legal guardian(s).

Exclusion Criteria:

1. Birth weight < 400 g or > 1,500 g.
2. Major apparent congenital abnormalities impacting cardio and pulmonary function identified before randomization, such as, but not limited to:

   * Clinically relevant Potter-like syndrome and any pulmonary congenital anomalies,
   * Clinically relevant congenital diaphragmatic hernia,
   * Omphalocele or gastroschisis, esophageal atresia,
   * Known or suspected cyanotic congenital heart disease (ie, tetralogy of fallot, transposition of the great arteries, etc).
3. Active do no resuscitate (DNR) order in place.
4. History of allergy or sensitivity to any surfactant or any component of zelpultide alfa.
5. Concurrent enrollment in any clinical study that utilizes treatments (investigational medical products or devices) outside of SOC or participation in studies within the last 30 days (or 5 half-lives of an IMP) prior to birth (for the mother) or up to week 36 PMA.
6. Any condition or situation that, in the Investigator's judgement, puts the neonate at significant risk, could confound the study results, or may interfere significantly with the neonate's participation in the study.

Ages: 0 Minutes to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 366 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2 or grade 3 Bronchopulmonary Dysplasia (BPD) or death | Week 36 Post Menstrual Age (PMA)
  BPD is defined and graded based on the classification according to Jensen et al., 2019 (2019 PMID: 30995069)

SECONDARY OUTCOMES:
Ventilator-free days | From birth to 36 weeks Post Menstrual Age (PMA)
  A ventilator-free day is defined as a natural calendar day without being on invasive mechanical ventilation (ie, invasive ventilation via ETT or tracheostomy); tracheostomy will be treated as all invasive ventilation.
Incidence of grade 2 or grade 3 Bronchopulmonary Dysplasia (BPD) | Week 36 Post Menstrual Age (PMA)
Incidence of death | Week 36 Post Menstrual Age (PMA)
Incidence of grade 2 or grade 3 Bronchopulmonary Dysplasia (BPD) or death assessed on 3 consecutive days at week 36 PMA | Week 36 Post Menstrual Age (PMA)
  BPD is defined and graded based on the classification according to Jensen et al., 2019 (2019 PMID: 30995069)
The proportion of subjects with no Bronchopulmonary Dysplasia (BPD), grade 1, grade 2, or grade 3 BPD | Week 36 Post Menstrual Age (PMA)
  BPD is defined and graded based on the classification according to Jensen et al., 2019 (2019 PMID: 30995069)
The proportion of subjects with no Bronchopulmonary Dysplasia (BPD), grade 1, grade 2, or grade 3 BPD assessed on 3 consecutive days at week 36 PMA | Week 36 Post Menstrual Age (PMA)
  BPD is defined and graded based on the classification according to Jensen et al., 2019 (2019 PMID: 30995069)
Ventilator-free days | From birth to day 28 of life
  A ventilator-free day is defined as a natural calendar day without being on invasive mechanical ventilation (ie, invasive ventilation via ETT or tracheostomy); tracheostomy will be treated as all invasive ventilation.
Total average days on supplemental oxygen | From birth to 36 Weeks Post Menstrual Age (PMA)
Total average days on continuous positive airway pressure (CPAP) or high flow nasal cannula (HFNC) | From birth to week 36 Post Menstrual Age (PMA)
Extubation rate | Study Day 7
Average preductal oxygen saturation measured by oxygen saturation to fraction of inspired oxygen ratio (SF) | From Study Days 1 to 7
Average preductal oxygen saturation measured by oxygen saturation index (OSI) | From Study Days 1 to 7
Incidence of grade 2 or grade 3 Bronchopulmonary Dysplasia (BPD) or death | Week 40 Post Menstrual Age (PMA)
  BPD is defined and graded based on the classification according to Jensen et al., 2019 (2019 PMID: 30995069)
Incidence of grade 2 or grade 3 Bronchopulmonary Dysplasia (BPD) | Week 40 Post Menstrual Age (PMA)
  BPD is defined and graded based on the classification according to Jensen et al., 2019 (2019 PMID: 30995069)
The proportion of subjects with no Bronchopulmonary Dysplasia (BPD), grade 1, grade 2, or grade 3 BPD | Week 40 Post Menstrual Age (PMA)
  BPD is defined and graded based on the classification according to Jensen et al., 2019 (2019 PMID: 30995069)
Incidence of grade 2 or grade 3 Bronchopulmonary Dysplasia (BPD) or death after excluding subjects with death at ≤ 14 days postnatal age | Week 36 and week 40 Post Menstrual Age (PMA)
  BPD is defined and graded based on the classification according to Jensen et al., 2019 (2019 PMID: 30995069)
Ventilator-free days | From birth to week 40 Post Menstrual Age (PMA)
  A ventilator-free day is defined as a natural calendar day without being on invasive mechanical ventilation (ie, invasive ventilation via ETT or tracheostomy); tracheostomy will be treated as all invasive ventilation.
Survival at 6, 12 and 24 months corrected age | 6, 12 and 24 month corrected age
Average number of hospitalizations and days in hospital | 6 and 12 months corrected age
Incidence of chronic respiratory morbidity | 12 month corrected age
Incidence of neurodevelopmental disability among survivors | 24 months corrected age
Severity and frequency of treatment-emergent adverse events (TEAEs) or treatment-emergent serious adverse events (TESAEs) | From start of treatment through week 36 Post Menstrual Age (PMA) or hospital discharge, whichever comes first
Immunogenicity analysis | Day 28 of life
  Determination of anti-SP-D antibodies in blood at day 28 of life compared to baseline), assessed in a subset of 60 patients

CONTACTS AND LOCATIONS:
Locations (20):
- Israel (3):
  - Bnai Zion Medical Center, Haifa
  - Shaare-Zedek Medical Center, Jerusalem
  - Ziv Medical Center, Safed
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale dei Bambini "V. Buzzi", Milan
  - Azienda Ospedale Università di Padova, Padua
- Spain (13):
  - Hospital General Universitario de Alicante Dr. Balmis, Alicante
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario Cruces - OSI Ezkerraldea-Enkarterri-Cruces, Bilbao
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No